CLINICAL TRIAL: NCT07038863
Title: Community Screening for Hepatitis B, C and Delta in the Mongolian Population Living in France
Brief Title: Community Screening and Management of Hepatitis B, C and Delta in the Mongolian Population Living in France
Acronym: Mondelta
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL24_0469; 2025-A00086-43 (Other: ID-RCB)
Record Dates: First submitted 2025-03-13; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HEPATITIS C (HCV); Hepatitis B Virus (HBV); Hepatitis D; Hepatocellular Carcinoma (HCC); Liver Fibrosis
Keywords: HBV; HCV; HDV; HCC
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Hepatitis D; Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening group (Experimental): This screening study focuses on Mongolian patients living in France. Screening will be organised in 11 centres in France, with 1 to 3 screening sessions per centre: patients will be informed of these screening sessions by the Mongolian Embassy in France, social networks and communities.
  Screening will be carried out by Rapid Diagnostic Orientation Test (TRODS) for hepatitis B (HBV), hepatitis C (HCV) and hepatitis B (HCV). If the TRODs are positive, a confirmatory serology test will be carried out, followed by specialist hepatology treatment.
  Interventions: Diagnostic Test: Community screening for hepatitis B, C and delta in the Mongolian population living in France

INTERVENTIONS:
Diagnostic Test: Community screening for hepatitis B, C and delta in the Mongolian population living in France — Screening will be organised in 11 centres in France, with 1 to 3 screening sessions per centre: patients will be informed of these screening sessions by the Mongolian Embassy in France, social networks and communities.
  During this screening visit, Rapid Diagnostic Orientation Test (RDOT) will be carried out to screen for HBV and HCV. If the RDOT is negative for both viruses, an information on transmission and prevention of viral infection will be given.
  If the RDOT is positive, confirmation of these tests by blood sampling will be organized and complementary biology (ASAT, ALAT, GGT, PAL, bilirubin total, bilirubin conjugated). If HBV RDOT positive, additional tubes will be collected for centralized analysis at the end of the study (VHD DNA, VHD genotyping, fibrotest and LCR1/2 test).
  Once these confirmatory tests have been carried out, the patient will be referred to a hepatology consultation.

SUMMARY:
In Mongolia, mortality from hepatocellular carcinoma (HCC) is one of the highest in the world. Viral hepatitis is the main cause of HCC: the prevalence of hepatitis B (HBV) estimated at 11% In Mongolia, hepatitis C (HCV) at 8.5%, and hepatitis Delta (HDV) at 40-60% in HBV-infected patients. Viral hepatitis are essentially asymptomatic and therefore require systematic screening for diagnosis. Once a diagnosis of chronic viral infection has been established, specific therapies are available to reduce the morbidity and mortality of these patients. A study carried out in California in the Mongolian community found an HBV prevalence of 9.7% and positive HDV serology in 41% of these patients.

There is a large Mongolian community in France, estimated at between 5,000 and 6,000 patients. Although the majority of these patients are covered by French social security; however, access to care and screening for viral hepatitis often remain difficult and insufficient for migrant or vulnerable populations in France The aim of this study is to screen the Mongolian community in France for viral hepatitis, and then initiate a program of care and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mongolian people
* Over 15 years of age
* Living in France
* Majors agree to participate or minors whose parental guardians agree to their child's participation in the study

Exclusion Criteria:

* People already followed for viral hepatitis, treated or not treated
* Persons deprived of their liberty by a judicial or administrative decision
* Adults subject to a legal protection measure (guardianship, curators)
* People participate in any interventional research except routine care research (old regulation) and category 2 research that does not interfere with the primary endpoint analysis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients positive for hepatitis B, hepatitis C and hepatitis D. | Visit 2 (Day 0 to Mounth 4)
  Number of patients with positive HBsAg (for HBV), positive serum HCV viral load (for HCV) and serum positive Delta viral load (for HDV) compared with all patients screened.

SECONDARY OUTCOMES:
Cascade of care for this screening strategy | 12 months after positive TROD screening
  Number of people tested positive for HBV, HCV or HDV who had a serological test, virological and elastometric evaluation, and hepatology consultation
Information on preventing viral hepatitis | Baseline
  Number of Mongolian people attending the information and prevention session offered on each screening day
Characterisation of liver fibrosis in patients with chronic viral hepatitis | Day 1 or up to 4 months
  Evaluation of hepatic fibrosis using biological test by FibroTest
Characterisation of liver fibrosis in patients with chronic viral hepatitis | Liver fibrosis will be assessed by elastometry and a FibroTest blood test, carried out according to the procedures of each centre, either during screening or at the specialist consultation.
  Evaluation of hepatic fibrosis using elastometry and biological test by FibroTest
Risk of hepatocellular carcinoma in patients positive for viral hepatitis | Day 1 or up to 4 months
  Evaluation of hepatocellular carcinoma (HCC) risk by biology (AFP)
Risk of hepatocellular carcinoma in patients positive for viral hepatitis | Day 1 or up to 4 months
  Evaluation of hepatocellular carcinoma (HCC) risk by liver imaging (ultrasound or CT (computed tomography) /MRI (magnetic resonance imaging))

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Expert Hépatites Virales Aquitaine, CHU de Bordeaux, Bordeaux
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor - Assistante Publique Hopitaux de Paris (APHP), Créteil
  - CHU Grenoble Alpes, Grenoble
  - CHRU Lille, Lille
  - Service d'Hépatologie, Institut d'hépatologie de Lyon, Hôpital Croix-Rousse, Hospices Civils de Lyon, Lyon
  - CHRU Rennes Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHRU Bretonneau, Tours